CLINICAL TRIAL: NCT05190874
Title: Grappler Interference Screw Post-Market Collection of Patient Reported Outcome Measures
Status: Completed | Type: Observational
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P41-SP-0002
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Ankle Injuries; Syndesmotic Injuries; Ankle Inversion Sprain; Deltoid Ankle Sprain; Achilles Tendon Rupture; Flexor Hallucis Longus on the Left; Flexor Hallucis Longus on the Right; Flexor Digitorum Longus on the Left; Flexor Digitorum Longus on the Right; Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Device: Grappler Interference Screw System: Foot and/or ankle procedure involving soft tissue attachment to bone using the Grappler Interference Screw System
  Interventions: Device: Grappler Interference Screw System

INTERVENTIONS:
Device: Grappler Interference Screw System — Foot and/or ankle procedure involving soft tissue attachment to bone using the Grappler® Interference Screw System

SUMMARY:
Ambispective, multi-surgeon, single site, consecutive case series to determine the safety, performance, and benefits of the Grappler(R) Interference Screw.

DETAILED DESCRIPTION:
This is an ambispective, multi-surgeon, single site, consecutive case series taking place in the United States. Once a subject is identified and informed consent is obtained from that subject, retrospective data will be collected from the subject's electronic medical record (EMR), and prospective data will be collected from subject-provided PROM's. A minimum of 16 and maximum of 23 subjects will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject underwent a foot and/or ankle procedure involving soft tissue attachment to bone using the Grappler Interference Screw System and completed by one of the designated investigators who are experienced in the use of such implants and the required specialized surgical techniques
* The subject signs a written informed consent form (ICF)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigational population will include a minimum of 23 subjects who have undergone a foot and/or ankle procedure that fulfill the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Device performance and benefits as related to Foot and Ankle Mobility Measure | 6 months post-operative
  Device performance and benefits as related to Foot and Ankle Mobility Measure Activities of Daily Living (0-84) and sports (0-32) subscales. The higher the score, the higher the level of function, with 100% representing no dysfunction.
Device performance and benefits as related to pain levels based on the Visual Analog Scale | 6 months post-operative
  Device performance and benefits as related to pain levels based on the Visual Analog Scale (range: 0 to 100; 0 = no pain; 100 = worst pain imaginable)of Daily Living (0-84) and sports (0-32) subscales. The higher the score, the higher the level of function, with 100% representing no dysfunction.
Device performance and benefits as related to pain levels based on Patient satisfaction | 6 months post-operative
  Device performance and benefits as related to patient satisfaction (very satisfied, good, fair, not satisfied)

SECONDARY OUTCOMES:
Safety will be assessed by recording the incidence of secondary procedures related to the index device | 6 months post-operative
  Safety will be assessed by recording the incidence of secondary procedures related to the index device

CONTACTS AND LOCATIONS:
Overall Officials: Jacy Legue, Study Director — Paragon 28
Locations (1):
- Orthopedic Foot and Ankle, Worthington, Ohio, United States

IPD SHARING:
Plan to Share IPD: No